CLINICAL TRIAL: NCT00299949
Title: Use of Whole Blood and Cell-rich Coagulation Assays for the Detection of Non-Overt DIC in Sepsis
Brief Title: Thrombin Generation and Thromboelastography in Non-overt DIC
Status: Terminated | Type: Observational
Why Stopped: Insufficient subject enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Deborah Brown, Associate Professor, Pediatrics, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-06-0012
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Sepsis; Disseminated Intravascular Coagulation
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be discarded after the study is completed.
Oversight: Data Monitoring Committee: No

SUMMARY:
Sepsis is the 13th most common cause of death in the United States, causing approximately 210,000 deaths per year. Once DIC has developed, irreversible organ injury has already occurred and the mortality rate is 70%. Inhibition of systemic coagulation with activated protein C concentrate has been the only therapy for sepsis introduced in the past several decades which has improved outcomes. Elucidation of the coagulopathic mechanisms early in the development of DIC may give rise to targeted therapies and strategies for early intervention. We hypothesize that an increase in endogenous thrombin potential precedes the development of overt DIC by a clinically significant time period. Our primary objective is to determine if endogenous thrombin potential (ETP) measured at first diagnosis of sepsis prior to the onset of DIC and organ failure is predictive of overt DIC and/or poor outcome. We will compare ETP to standard coagulation assays and the clinical assessment of DIC using the ISTH criteria for overt DIC. A secondary objective of this study is to determine if host coagulation variables predispose to the development of DIC and poor clinical outcome during sepsis.

DETAILED DESCRIPTION:
Activation of the coagulation system occurs early in patients with sepsis, although clinically overt disseminated intravascular coagulation (DIC) is identified in only a minority of patients with severe sepsis. Uncontrolled activation of the coagulation system may contribute to the pathophysiology of multiple organ failure and the subsequent morbidity and mortality of sepsis. Identification of risk factors predicting progression to severe sepsis and DIC has been elusive. We propose that whole blood and cell-rich coagulation assays will offer improved sensitivity to both the procoagulant and anti-coagulant changes which occur early in sepsis and will improve recognition of non-overt DIC. Future studies will address whether these assays have sufficiently high predictive value to identify subgroups of patients who could benefit from early intervention.

Specific Aims:

1. We hypothesize that increased thrombin generation will precede development of overt DIC by a clinically significant time period. Our primary objective is to determine if endogenous thrombin potential measured at first diagnosis of sepsis prior to the onset of DIC and organ failure is predictive of overt DIC.
2. There is significant individual variation among the healthy population in endogenous thrombin generation due to known and unknown polymorphisms within coagulation proteins. We predict that host variables in thrombin generation will contribute to susceptibility to DIC and poor outcome during sepsis. A secondary objective of this study is to determine if host coagulation variables predispose to the morbidity and mortality associated with sepsis.

Experimental Design and Methods

The study design will be a prospective observational study of patients presenting to the Memorial Hermann Hospital Emergency Department with sepsis. Criteria for sepsis include evidence of systemic inflammatory response syndrome as defined by the ACCP/SCCM Consensus Conference, and a known or suspected infection. Exclusion criteria include signs of severe sepsis or septic shock, as defined by the ACCP/SCCM Consensus Conference, at presentation, including: organ dysfunction, hypoperfusion and perfusion abnormalities. Chronic medical conditions associated with immune suppression or coagulopathies, such as neutropenia and sickle cell disease, and use of medications leading to immune dysfunction or coagulopathies, such as chronic steroid use or anti-coagulation will also be reasons for exclusion. In addition, because of the volume of blood required from each patient for laboratory studies, only patients 25 kg body weight or more will be enrolled. Withdrawal from the study will be at the discretion of the treating physician or subject. All efforts will be made to collect clinical information from patients who have withdrawn.

Inclusion criteria

* Known or suspected infection as determined by the treating physician Patient to be admitted to the hospital
* Systemic Inflammatory Response Syndrome: 3 of the following 4 criteria:
* Temperature > 38 C or < 35 C
* Heart rate > 90 beats/min, except in patients with a medical condition known to increase the heart rate or those receiving treatment that would prevent tachycardia.
* Respiratory rate > 20 breaths/min or PaC02 < 32 mmHg, or on mechanical ventilation for an acute respiratory process.
* White blood cell count > 12,000/mm3, < 4,000/mm3, or > 10% bands

Exclusion criteria

* - Use of the following medications: unfractionated heparin to treat an active thrombotic event within 8 hours before the infusion; low-molecular-weight heparin at a higher dose than recommended for prophylactic use within 12 hours before the infusion, warfarin used within 7 days of study entry, aspirin use at a dose of more than 650 mg/day within 3 days before the study, thrombolytic therapy within 3 days before the study, glycoprotein IIb/IIIa antagonists within 7 days before the study entry, administration of activated protein C (Xigris ) in the 24 hours before study entry.
* Neutropenia
* Hemophilia
* Diabetic ketoacidosis
* Weight < 25 kg

Patients will be enrolled in the emergency department within 2 hours of meeting eligibility. Written informed consent will be obtained from the patients or their authorized representatives. Blood samples will be collected by peripheral venipuncture during the first hour after enrollment and then once daily for 7 days (see Appendix A).

Patients will be withdrawn from the study if blood sampling is not performed within 2 hours of obtaining informed consent.

Clinical data collection Clinical data forms (see Appendix B) will be completed at the time of enrollment and daily for 7 days , at hospital discharge, and at 28 days. Clinicians will be blinded to the results of the research laboratory tests.

Laboratory Methods

Blood and plasma Each patient will have 15 ml blood collected at enrollment. Specimens will be obtained through antecubital venipuncture. Free flow or minimal suction will be employed; vacuum containers will be avoided. Specimens for platelet-poor plasma (PPP) and whole blood analysis will be collected into siliconized glass tubes with 0.105M tri-sodium citrate in the ratio of 1 part anticoagulant to 9 parts whole blood. PPP will be separated within 60 minutes and analyzed immediately. Platelet-rich plasma (PRP) specimens will be separated from the upper ¾ volume of plasma supernatant after centrifugation at 265g for 10 minutes at room temperature. The platelets will be counted on a Beckman Coulter counter and adjusted to 150 X 109 platelets/l with autologous PPP. PRP will be used within 60 minutes. Cbc, PT/PTT, Fibrinogen, d-dimer, Protein C activity, Protein S activity, ATIII activity, Factor V Leiden mutation, Prothrombin G20210A mutation analysis will be performed in Memorial Herman Hospital clinical laboratories.

RoTEG

Whole blood specimens will be drawn as described above. Measurements will be performed on two roTEG Coagulation Analyzers from Pentapharm. RoTEG all-plastic reaction cups are procured from the manufacturer. Polypropylene and polyethylene pipettes are used to handle reagents and blood. Citrated whole blood will be re-calcified by 20 mcl 0.2 mol/L CaCl2 and activated by 20 mcl solution of recombinant human TF (Innovin) diluted 1:1000 using a sodium barbital buffer. The measured parameters have been defined by the manufacturer as follows: The clotting time(CT) is the time in seconds from Ca2+ activation of coagulation and until an increase in elasticity corresponding to 2 graphical mm is obtained on the ordinate. The clot formation time (CFT) is the time in seconds passing while the elasticity increases from 2 mm to 20 mm on the ordinate. The maximum clot formation (MCF) expresses the maximum strength in millimeters of the final clot. Several additional parameters representing the continuous registration of clot formation have been defined by Sorensen et al 28: the maximum velocity (MaxVel) of clot formation, the time to maximum velocity (T,MaxVel) of clot formation, and the area under the velocity curve (AUC).

Thrombin Generation

Calibrated automated thrombin generation measurements will be performed using the Hemker methodology. 29 Platelet rich plasma (PRP) will be prepared as described above. Fluorogenic substrate and chromogenic thrombin will be purchased through Thermolabsystems, and recombinant relipidated tissue factor(TF) through Dade Behring. alpha 2 macroglobulin-thrombin complex used as a calibrator will be purchased through Thrombolabsystems. The thrombograms will be measured in a 96-well plate fluorometer (Ascent reader, Thrombolabsystems) and analyzed with software purchased through Thrombinoscope. Experiments will be carried out in quadruplicate and compared to a calibrator. To each well 80 mcl of plasma will be added, followed by the calibrator or buffer, then the "trigger": 20 mcl of 3 mM of TF. The plate will be placed in the fluorometer and allowed to warm to 37 C. The instrument dispenses 20 mcl of Fluorogenic substrate 2.5 mM and CaCl2 100 mM (FluCa) to all the wells to be measured, registers this as zero time, shakes them for 10 s and starts reading. During the measurement, the program compares the readings from the TG and the CL, calculates thrombin concentration and displays the thrombin concentration in time. The peak thrombin is the highest thrombin concentration reached during the time course of thrombin formation and inhibition. The thrombin potential is the amount of thrombin that is formed within 60 minutes (Area under the curve). The lag phase and the peak time refer to the start and velocity of thrombin formation, respectively.

Data Management Data will be collected on paper forms which will be designed by the GCRC informatics core section. The GCRC informatics core will maintain data on a secure database (Access). Each subject will be assigned a unique ID reflecting the order in which enrollment took place.

Data Analysis and Presentation

This is a pilot study intended to provide the preliminary data for future clinical studies. Descriptive statistics will be used to characterize ETP and roTEG at initial presentation of sepsis. Means and ranges will be reported for each of the variables in the thrombin generation assay (lag time, slope of rise, peak value, and area under the curve) and roTEG (Clot formation time (CFT), maximum clot formation (MCF), maximum velocity (MaxVel) of clot formation, time to maximum velocity (T,MaxVel) of clot formation, and area under the velocity curve (AUC)). The primary objective of this study is to compare ETP at presentation to the development of DIC, as defined by a positive ISTH DIC score. The secondary objective will be to compare host coagulation variables, including ETP, roTEG, Pro C, Pro S, ATIII, FVL, and prothrombin G20210A mutation at presentation, with the secondary outcome measures of 28-day mortality and organ dysfunction. All statistics will be performed using NCSS/PASS.

Sample size determination: There are no published reports of thrombin generation assays or thromboelastography in sepsis, or DIC. In our previous studies of patients taking an anticoagulant (warfarin), there was a 400% decrement of ETP (1719 to 404). In order to derive a mean ETP with a target width of 100 and 95% confidence interval, assuming a standard deviation of 259, we will need to enroll 100 patients.

We will employ the following statistical methods for the analysis of data:

Specific Aim #1: The endogenous thrombin potential (ETP) is the area under the curve of the thrombin generation assay. The values are continuous and range from 0 to 2,500. Maximum clot formation (MCF) from the roTEG will also be used to approximate ETP. The DIC score will be calculated and coded as a dichotomous variable: Yes (score > 5) or No (score < 5). A receiver operating curve will be derived for ETP and MCT and its sensitivity and specificity for predicting DIC. If the area under the curve is found to be significant, an optimal cut-off value with the highest degree of accuracy will be chosen. This value will be used to estimate the predictive value of the test. Positive predictive value will be calculated with the formula: # patients with ETP or MCT above the cut-off and development of DIC / # patients with positive DIC score. The predictive value of a negative DIC score will be calculated using the formula: # patients with ETP or MCT below the cut-off and no progression to DIC / # patients with negative DIC score.

Specific Aim #2: A multivariate analysis will be done to determine which of the predictor variables (ETP, MCT, Pro C, Pro S, ATIII, FVL, ProG20210A, DIC) are associated with the secondary dichotomous outcome measures: organ dysfunction at 28 days (Any/None), 28-day mortality (Dead/Alive).

ELIGIBILITY:
Inclusion Criteria:

* Systemic inflammatory response syndrome with known or suspected infection
* Patient to be admitted to the hospital

Exclusion Criteria:

* Diabetic ketoacidosis, Hemophilia, weight < 25 kg, use of hemostatic agents prior to entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients arriving in Emergency Department with sepsis (systemic inflammatory response syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  ETP will be used to predict 28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Brown, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States